CLINICAL TRIAL: NCT06676709
Title: Effect of IMMUNEPOTENT-CRP, a Bovine Dialyzable Leukocyte Extract, on Serum Pro-Inflammatory Cytokines in Outpatients with Mild to Moderate COVID-19: a Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: Effect of IMMUNEPOTENT-CRP on Serum Pro-Inflammatory Cytokines in Mild to Moderate COVID-19
Acronym: ICRPDLECOVID
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Collaborators: Laboratorio de Inmunologia y Virologia - UANL (Other); Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Dr. Jose Manuel Vazquez-Guillen, Full-Time Research Professor, Universidad Autonoma de Nuevo Leon
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EN21-00050/LIVFCB-2021-001; EN21-00050 (Other: Universidad Autónoma de Nuevo León)
Record Dates: First submitted 2024-10-29; First posted 2024-11-06 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: COVID-19; SARS-CoV2 Infection
Keywords: Cytokine storm; Mild to moderate COVID-19; Inflammatory cytokines; Dialyzable Leukocyte Extract (DLE); IMMUNEPOTENT-CRP (I-CRP)
MeSH Terms: conditions — COVID-19; Cytokine Release Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- I-CRP group (Experimental): IMMUNEPOTENT-CRP (I-CRP) was supplied in a 5 Unit (U) per vial presentation. One U is defined as the lyophilized product obtained from the dialysis of 1×10^8 bovine spleen cells. The dosing schedule extended over 14 days. On the first day (Day 0), outpatients ingested seven doses at two-hour intervals each one. From days one through four, four doses were taken one every four hours, and from days five to thirteen, three doses were consumed one every eight hours.
  Interventions: Biological: IMMUNEPOTENT-CRP (I-CRP)
- Placebo control (Placebo Comparator): The placebo was prepared from a lyophilized corn starch extract and was provided in an identical appearance and presentation to IMMUNEPOTENT-CRP (I-CRP). The dosing schedule extended over 14 days. On the first day (Day 0), outpatients ingested seven doses at two-hour intervals each one. From days one through four, four doses were taken one every four hours, and from days five to thirteen, three doses were consumed one every eight hours.
  Interventions: Biological: Placebo Comparator

INTERVENTIONS:
Biological: IMMUNEPOTENT-CRP (I-CRP) — IMMUNEPOTENT-CRP (I-CRP), a bovine dialyzable leukocyte extract (DLE) obtained from disrupted spleen cells, is a mixture of low-molecular-weight peptides (<12 kDa) that exhibit non-specific immunomodulatory properties.
  Other Names: Bovine Dialyzable Leukocyte Extract (DLE)
  Arms: I-CRP group
Biological: Placebo Comparator — The placebo was prepared from a lyophilized corn starch extract and was provided in an identical appearance and presentation to IMMUNEPOTENT-CRP (I-CRP).
  Arms: Placebo control

SUMMARY:
In this study, the effects of IMMUNEPOTENT-CRP (I-CRP), a dialyzable leukocyte extract (DLE) derived from bovine spleen cells, on the levels of key inflammatory cytokines in outpatients with COVID-19 were examined. I-CRP has been previously studied for its ability to regulate the immune system in other conditions, such as cancer and sepsis. Based on its potential to reduce harmful inflammation, the study aimed to determine if similar benefits could be observed in COVID-19 outpatients.

DETAILED DESCRIPTION:
Outpatients with mild to moderate COVID-19 symptoms and a confirmed SARS-CoV-2 infection were enrolled. These patients were randomly assigned to receive either IMMUNEPOTENT-CRP (I-CRP) or a placebo over a 14-day period. The study was double-blind, meaning neither the patients nor the researchers knew who was receiving I-CRP or placebo, ensuring unbiased results. The main objective of the study was to measure changes in the levels of specific cytokines and chemokines in the blood-IL-1β, IL-6, IL-10, TNF-α, IFN-α, IFN-γ, and IL-8-which are key players in the inflammatory response linked to severe COVID-19 cases. High levels of these molecules are associated with worse outcomes and more severe symptoms. Additionally, other markers of inflammation and immune system activity, such as lactate dehydrogenase (LDH), high-sensitivity C-reactive protein (hs-CRP), ferritin, and D-dimer, were measured, as these are commonly used to assess the severity of inflammation and risk of complications in COVID-19 patients.

Throughout the study, outpatients were regularly monitored for symptoms, and their vital signs-such as oxygen levels and body temperature-were checked during home visits. Blood samples were collected at different intervals to measure cytokine levels and the other included inflammatory markers. Patients were also tested four times for the presence of the virus to determine their infection status during the follow-up period.

ELIGIBILITY:
Outpatients Inclusion Criteria:

* Laboratory-confirmed SARS-CoV-2 infection (by antigen or RT-qPCR test).
* With mild to moderate symptoms of COVID-19.
* Aged ≥ 18 years.
* Not participating in any other clinical study.
* Written informed consent duly signed.

Outpatients Exclusion Criteria:

* Undergoing any process of primary or secondary immunosuppression.
* Any autoimmune disease.
* Receiving chemotherapy.
* History of lymphoma or any malignancy.
* Pregnancy or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-03-05 (Actual)

PRIMARY OUTCOMES:
Cytokine and Chemokine Serum Levels Evaluation | Assessments were performed at baseline (Day 0), and during the intervention period at Day 7 and Day 14.
  Serum levels of IL-1β, IL-6, IL-10, TNF-α, IFN-α, IFN-γ, and IL-8 were measured using the Human Cytokine/Chemokine Magnetic Bead Panel (Milliplex, Darmstadt, Germany). Cytokine and chemokine concentrations in the serum are expressed in pg/mL.

SECONDARY OUTCOMES:
Lactate Dehydrogenase (LDH) Levels | Measurements were taken at baseline (Day 0), Day 7, and Day 14 during the intervention period.
  Plasma levels of lactate dehydrogenase (LDH) were measured using standard biochemistry tests. Reference normal values are 230-460 mg/dL.
High-Sensitivity C-Reactive Protein (hs-CRP) Levels | Measurements were taken at baseline (Day 0), Day 7, and Day 14 during the intervention period.
  Serum levels of high-sensitivity C-reactive protein (hs-CRP) were measured using standard biochemistry tests. Reference normal values are 0.0-0.3 mg/dL.
Ferritin Levels | Measurements were taken at baseline (Day 0), Day 7, and Day 14 during the intervention period.
  Serum levels of ferritin were measured using standard biochemistry tests. Reference normal values are 13-150 ng/mL.
D-Dimer Levels | Measurements were taken at baseline (Day 0), Day 7, and Day 14 during the intervention period.
  Plasma levels of D-dimer were measured using standard biochemistry tests. Reference normal values are 0.0-0.5 μg/mL.
Lymphocyte Subpopulations | Lymphocyte subpopulation counts in whole blood were measured at baseline (Day 0), Day 7, and Day 14 during the administration of I-CRP or placebo.
  The percentages (%) of lymphocyte subpopulations in whole blood were determined using the BD Multitest 6-color TBNK reagent kit (BD Biosciences, San Jose, USA) and analyzed with the BD FACSCanto™ flow cytometer (BD Biosciences).
SARS-CoV-2 Infection Status Evaluation | SARS-CoV-2 infection status was evaluated at baseline (Day 0), Day 7, Day 14, and Day 30 during outpatient follow-up.
  Nasopharyngeal/oropharyngeal (NP/OP) flocked swabs collected in 3-5 mL of viral transport medium (VTM) were used to determine SARS-CoV-2 infection status via RT-qPCR. The 2019-nCoV CDC EUA Kit (IDT, Coralville, USA) primers and probe set were used for the assay. RT-qPCR results with a sigmoidal amplification curve and a cycle threshold (Ct) value of ≤37 were considered positive for SARS-CoV-2, while Ct values of 38 and above were considered negative.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Rodriguez-Padilla, Ph.D., Study Director — Universidad Autonoma de Nuevo Leon; Rene Rodriguez-Gutierrez, Ph.D., Study Chair — Universidad Autonoma de Nuevo Leon; Jose Manuel Vazquez-Guillen, Ph.D., Principal Investigator — Universidad Autonoma de Nuevo Leon
Locations (2):
- Mexico (2):
  - Hospital Universitario "Dr. Jose E. Gonzalez", Universidad Autonoma de Nuevo Leon, Monterrey, Nuevo León
  - Laboratorio de Inmunologia y Virologia, San Nicolás de los Garza, Nuevo León

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) to be shared with other researchers will include the following variables related to the study participants:
  * Basic demographic information (such age, sex, and others)
  * Serum levels of pro-inflammatory cytokines
  * Relevant clinical data related to SARS-CoV-2 infection, such as symptom severity and clinical progression
  * Data on treatment group allocation (IMMUNEPOTENT-CRP or placebo)
  Prior to sharing the data, all identifiable participant information will be anonymized to ensure privacy and confidentiality. Measures will be taken to prevent any possible re-identification of participants.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data will be available for a period of 3 years following the publication of the study.
Access Criteria: The IPD will be made available to other researchers after the publication of the study results in a peer-reviewed scientific journal. Data will be available upon reasonable request and subject to approval by the study's Ethics Committee. Interested researchers may request access to the IPD by contacting the principal investigator of the study. Requests must include a clear description of the research purpose, and researchers must agree to use the data only for the specified purposes and comply with applicable ethical and data protection regulations.

REFERENCES:
- [Background] Franco-Molina MA, Santana-Krímskaya SE, Zarate-Triviño DG, Zapata-Benavides P, Hernández-Martínez SP, Cervantes-Wong F, et al. Bovine dialyzable leukocyte extract immunepotent CRP: Evaluation of biological activity of the modified product. Appl Sci 2021;11. https://doi.org/10.3390/app11083505.
- [Background] Ayala MC, Gonzalez NM, Palacios G, Rivera-Morales LG, Rodriguez-Padilla C. [Dialyzed leukocyte extracts for the treatment of recurrent and severe infections in pediatric patients with cellular immunodeficiency: 15 years of experience]. Rev Alerg Mex. 2019 Jan-Mar;66(1):27-37. doi: 10.29262/ram.v66i1.531. Spanish. PMID 31013404
- [Background] Franco-Molina MA, Mendoza-Gamboa E, Castillo-Leon L, Tamez-Guerra RS, Rodriguez-Padilla C. Bovine dialyzable leukocyte extract protects against LPS-induced, murine endotoxic shock. Int Immunopharmacol. 2004 Dec 15;4(13):1577-86. doi: 10.1016/j.intimp.2004.06.014. PMID 15454111
- [Background] Armides Franco-Molina M, Mendoza-Gamboa E, Castillo-Tello P, Tamez-Guerra RS, Villarreal-Trevino L, Tijerina-Menchaca R, Castillo-Leon L, Zapata-Benavides P, Rodriguez-Padilla C. In vitro antibacterial activity of bovine dialyzable leukocyte extract. Immunopharmacol Immunotoxicol. 2006;28(3):471-83. doi: 10.1080/08923970600928072. PMID 16997795
- [Background] Franco-Molina MA, Mendoza-Gamboa E, Miranda-Hernandez D, Zapata-Benavides P, Castillo-Leon L, Isaza-Brando C, Tamez-Guerra RS, Rodriguez-Padilla C. In vitro effects of bovine dialyzable leukocyte extract (bDLE) in cancer cells. Cytotherapy. 2006;8(4):408-14. doi: 10.1080/14653240600847266. PMID 16923617
- [Background] Mendoza-Gamboa E, Franco-Molina MA, Zapata-Benavides P, Castillo-Tello P, Vera-Garcia ME, Tamez-Guerra RS, Rodriguez-Padilla C. Bovine dialyzable leukocyte extract modulates AP-1 DNA-binding activity and nuclear transcription factor expression in MCF-7 breast cancer cells. Cytotherapy. 2008;10(2):212-9. doi: 10.1080/14653240801891659. PMID 18368600
- [Background] Franco-Molina MA, Mendoza-Gamboa E, Zapata-Benavides P, Castillo-Tello P, Isaza-Brando CE, Zamora-Avila D, Rivera-Morales LG, Miranda-Hernandez DF, Sierra-Rivera CA, Vera-Garcia ME, Tamez-Guerra RS, Rodriguez-Padilla C. Antiangiogenic and antitumor effects of IMMUNEPOTENT CRP in murine melanoma. Immunopharmacol Immunotoxicol. 2010 Dec;32(4):637-46. doi: 10.3109/08923971003663253. Epub 2010 Mar 5. PMID 20205507
- [Background] Lara HH, Ixtepan-Turrent L, Garza-Trevino EN, Badillo-Almaraz JI, Rodriguez-Padilla C. Antiviral mode of action of bovine dialyzable leukocyte extract against human immunodeficiency virus type 1 infection. BMC Res Notes. 2011 Nov 1;4:474. doi: 10.1186/1756-0500-4-474. PMID 22044844
- [Background] Sierra-Rivera CA, Franco-Molina MA, Mendoza-Gamboa E, Zapata-Benavides P, Santaolalla-Tapia J, Coronado-Cerda EE, Tamez-Guerra RS, Rodriguez-Padilla C. Effect of bovine dialyzable leukocyte extract on induction of cell differentiation and death in K562 human chronic myelogenous leukemia cells. Oncol Lett. 2016 Dec;12(6):4449-4460. doi: 10.3892/ol.2016.5285. Epub 2016 Oct 18. PMID 28101208
- [Background] Lorenzo-Anota HY, Reyes-Ruiz A, Calvillo-Rodriguez KM, Mendoza-Reveles R, Urdaneta-Peinado AP, Alvarez-Valadez KM, Martinez-Torres AC, Rodriguez-Padilla C. IMMUNEPOTENT CRP increases intracellular calcium through ER-calcium channels, leading to ROS production and cell death in breast cancer and leukemic cell lines. EXCLI J. 2023 Mar 16;22:352-366. doi: 10.17179/excli2022-5568. eCollection 2023. PMID 37223080
- [Background] Garcia Coronado PL, Franco Molina MA, Zarate Trivino DG, Menchaca Arredondo JL, Zapata Benavides P, Rodriguez Padilla C. Putative Wound Healing Induction Functions of Exosomes Isolated from IMMUNEPOTENT CRP. Int J Mol Sci. 2023 May 18;24(10):8971. doi: 10.3390/ijms24108971. PMID 37240318
- [Background] Calvillo-Rodriguez KM, Lorenzo-Anota HY, Rodriguez-Padilla C, Martinez-Torres AC, Scott-Algara D. Immunotherapies inducing immunogenic cell death in cancer: insight of the innate immune system. Front Immunol. 2023 Nov 23;14:1294434. doi: 10.3389/fimmu.2023.1294434. eCollection 2023. PMID 38077402
- [Background] Coronado-Cerda EE, Franco-Molina MA, Mendoza-Gamboa E, Prado-Garcia H, Rivera-Morales LG, Zapata-Benavides P, Rodriguez-Salazar Mdel C, Caballero-Hernandez D, Tamez-Guerra RS, Rodriguez-Padilla C. In Vivo Chemoprotective Activity of Bovine Dialyzable Leukocyte Extract in Mouse Bone Marrow Cells against Damage Induced by 5-Fluorouracil. J Immunol Res. 2016;2016:6942321. doi: 10.1155/2016/6942321. Epub 2016 Apr 17. PMID 27191003
- [Background] Rodriguez-Salazar MDC, Franco-Molina MA, Mendoza-Gamboa E, Martinez-Torres AC, Zapata-Benavides P, Lopez-Gonzalez JS, Coronado-Cerda EE, Alcocer-Gonzalez JM, Tamez-Guerra RS, Rodriguez-Padilla C. The novel immunomodulator IMMUNEPOTENT CRP combined with chemotherapy agent increased the rate of immunogenic cell death and prevented melanoma growth. Oncol Lett. 2017 Jul;14(1):844-852. doi: 10.3892/ol.2017.6202. Epub 2017 May 18. PMID 28693241
- [Background] Martinez-Torres AC, Reyes-Ruiz A, Benitez-Londono M, Franco-Molina MA, Rodriguez-Padilla C. IMMUNEPOTENT CRP induces cell cycle arrest and caspase-independent regulated cell death in HeLa cells through reactive oxygen species production. BMC Cancer. 2018 Jan 3;18(1):13. doi: 10.1186/s12885-017-3954-5. PMID 29298674
- [Background] Martinez-Torres AC, Gomez-Morales L, Martinez-Loria AB, Uscanga-Palomeque AC, Vazquez-Guillen JM, Rodriguez-Padilla C. Cytotoxic activity of IMMUNEPOTENT CRP against non-small cell lung cancer cell lines. PeerJ. 2019 Sep 27;7:e7759. doi: 10.7717/peerj.7759. eCollection 2019. PMID 31579619
- [Background] Santana-Krimskaya SE, Franco-Molina MA, Zarate-Trivino DG, Prado-Garcia H, Zapata-Benavides P, Torres-Del-Muro F, Rodriguez-Padilla C. IMMUNEPOTENT CRP plus doxorubicin/cyclophosphamide chemotherapy remodel the tumor microenvironment in an air pouch triple-negative breast cancer murine model. Biomed Pharmacother. 2020 Jun;126:110062. doi: 10.1016/j.biopha.2020.110062. Epub 2020 Mar 12. PMID 32172064
- [Background] Lorenzo-Anota HY, Martinez-Torres AC, Scott-Algara D, Tamez-Guerra RS, Rodriguez-Padilla C. Bovine Dialyzable Leukocyte Extract IMMUNEPOTENT-CRP Induces Selective ROS-Dependent Apoptosis in T-Acute Lymphoblastic Leukemia Cell Lines. J Oncol. 2020 Jun 8;2020:1598503. doi: 10.1155/2020/1598503. eCollection 2020. PMID 32587616
- [Background] Martinez-Torres AC, Reyes-Ruiz A, Calvillo-Rodriguez KM, Alvarez-Valadez KM, Uscanga-Palomeque AC, Tamez-Guerra RS, Rodriguez-Padilla C. IMMUNEPOTENT CRP induces DAMPS release and ROS-dependent autophagosome formation in HeLa and MCF-7 cells. BMC Cancer. 2020 Jul 13;20(1):647. doi: 10.1186/s12885-020-07124-5. PMID 32660440
- [Background] Lorenzo-Anota HY, Martinez-Loria AB, Tamez-Guerra RS, Scott-Algara D, Martinez-Torres AC, Rodriguez-Padilla C. Changes in the natural killer cell repertoire and function induced by the cancer immune adjuvant candidate IMMUNEPOTENT-CRP. Cell Immunol. 2022 Apr;374:104511. doi: 10.1016/j.cellimm.2022.104511. Epub 2022 Mar 26. PMID 35381435
- [Background] Rivera-Lazarin AL, Martinez-Torres AC, de la Hoz-Camacho R, Guzman-Aguillon OL, Franco-Molinaa MA, Rodriguez-Padilla C. The bovine dialyzable leukocyte extract, immunepotent CRP, synergically enhances cyclophosphamide-induced breast cancer cell death, through a caspase-independent mechanism. EXCLI J. 2023 Jan 13;22:131-145. doi: 10.17179/excli2022-5389. eCollection 2023. PMID 36998710
- [Background] Rivera-Lazarin AL, Calvillo-Rodriguez KM, Izaguirre-Rodriguez M, Vazquez-Guillen JM, Martinez-Torres AC, Rodriguez-Padilla C. Synergistic Enhancement of Chemotherapy-Induced Cell Death and Antitumor Efficacy against Tumoral T-Cell Lymphoblasts by IMMUNEPOTENT CRP. Int J Mol Sci. 2024 Jul 20;25(14):7938. doi: 10.3390/ijms25147938. PMID 39063180
- [Background] Lara HH, Turrent LI, Garza-Trevino EN, Tamez-Guerra R, Rodriguez-Padilla C. Clinical and immunological assessment in breast cancer patients receiving anticancer therapy and bovine dialyzable leukocyte extract as an adjuvant. Exp Ther Med. 2010 May;1(3):425-431. doi: 10.3892/etm_00000066. Epub 2010 May 1. PMID 22993557
- [Background] Franco-Molina MA, Mendoza-Gamboa E, Castillo-Tello P, Isaza-Brando CE, Garcia ME, Castillo-Leon L, Tamez-Guerra RS, Rodriguez-Padilla C. Bovine dialyzable leukocyte extract modulates cytokines and nitric oxide production in lipopolysaccharide-stimulated human blood cells. Cytotherapy. 2007;9(4):379-85. doi: 10.1080/14653240701320262. PMID 17573613
- [Background] Franco-Molina MA, Mendoza-Gamboa E, Castillo-Leon L, Tamez-Guerra RS, Rodriguez-Padilla C. Bovine dialyzable leukocyte extract modulates the nitric oxide and pro-inflammatory cytokine production in lipopolysaccharide-stimulated murine peritoneal macrophages in vitro. J Med Food. 2005 Spring;8(1):20-6. doi: 10.1089/jmf.2005.8.20. PMID 15857204
- [Background] Franco-Molina MA, Mendoza-Gamboa E, Zapata-Benavides P, Vera-Garcia ME, Castillo-Tello P, Garcia de la Fuente A, Mendoza RD, Garza RG, Tamez-Guerra RS, Rodriguez-Padilla C. IMMUNEPOTENT CRP (bovine dialyzable leukocyte extract) adjuvant immunotherapy: a phase I study in non-small cell lung cancer patients. Cytotherapy. 2008;10(5):490-6. doi: 10.1080/14653240802165681. PMID 18821359
- [Background] Reyes-Ruiz A, Calvillo-Rodriguez KM, Martinez-Torres AC, Rodriguez-Padilla C. The bovine dialysable leukocyte extract IMMUNEPOTENT CRP induces immunogenic cell death in breast cancer cells leading to long-term antitumour memory. Br J Cancer. 2021 Apr;124(8):1398-1410. doi: 10.1038/s41416-020-01256-y. Epub 2021 Feb 3. PMID 33531687